CLINICAL TRIAL: NCT04213417
Title: Effectiveness of Combining Matrix Rhythm Therapy and Bobath Toncept on Increased Muscle Tone, Balance and Gait Parameters in Stroke Individuals With Spastic Hemiparesis: A Single-Blind, Randomized, Controlled Clinical Trial
Brief Title: Effectiveness of Matrix Rhythm Therapy on Increased Muscle Tone, Balance and Gait Parameters in Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, AYŞE ÜNAL, Research assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27.12.2016/81261
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Stroke
Keywords: stroke survivor; spasticity; Matrix Rhythm Therapy; balance; gait
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bobath therapy plus Matrix Rhythm Therapy (Experimental): MRT application that was applied to the study group in addition to the Bobath therapy was applied to the affected side of the body and lower extremity for 60 minutes in each session.
  Interventions: Other: Bobath therapy and Matrix Rhythm Therapy
- Bobath therapy (Active Comparator): Both groups were treated with the Bobath therapy as a neurodevelopmental therapy.
  Interventions: Other: Bobath therapy

INTERVENTIONS:
Other: Bobath therapy and Matrix Rhythm Therapy — MRT application that was applied to the study group in addition to the BC was applied to the affected side of the body and lower extremity for 60 minutes in each session.The treatment was started from the thoracic region and a treatment direction was toward the lower extremity in the affected side.During the MRT procedure, the patient's active participation was ensured and the treatment was combined with the exercises.The patients were informed about MRT verbally and in writing before the application. Participants were treated 3 days a week for 4 weeks for a total of 12 sessions.
  Arms: Bobath therapy plus Matrix Rhythm Therapy
Other: Bobath therapy — Both groups were treated with the BC as a neurodevelopmental therapy. Considering individual requirements and wishes of the patient, an exercise program that supports active participation of the person was established.Each treatment session was performed for 60 minutes.The treatment program that was established appropriately according to the patient contained weight transfer to the affected side in different positions,approximation to increase proprioceptive input, providing sensorial input to the sole of the foot using materials such as sensory ball,foot-ankle mobilization,functional reach activities, forward-side step, gait, and balance activities. Participants in both groups were treated 3 days a week for 4 weeks for a total of 12 sessions.
  Arms: Bobath therapy

SUMMARY:
Matrix-Rhythm-Therapy(MRT) has been included in neuro-rehabilitation program for stroke patients to regulate increased muscle tone.

There are no controlled studies with large sample size on the efficacy of MRT on spasticity. In this context,to the best of our knowledge, our study is the first study on this subject. The results of the study will develop a new perspective for management of spasticity and will ensure more common use of MRT.Further studies are needed on superiority of MRI over other treatment methods used in gait and balance rehabilitation of hemiparetic individuals. The aim of this study was to investigate the effectiveness of combining Bobath therapy (BT) and MRT on muscle tone,balance and gait parameters in stroke individuals with spastic hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* aged between
* to discharge from the hospital,
* to have single-sided hemiparesis for the first time,
* to have hemiparesis at least four weeks earlier.
* to have Modified Rankin Score of ≤3, Modified Ashworth Scale score between 1-5 for the lower extremity.

Exclusion Criteria:

* to use a cardiac pacemaker,
* to have aphasia, open wound in the area to be treated,
* to have circulatory problem, skin lesions, other neurological, psychiatric and/or orthopedic problems other than hemiparesis affecting gait.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 20-65 years
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 1 year
  In 1987, Bohannon et al. developed the MAS(0,1,1+,2,3,4). In various studies, "0,1,2,3,4,5"scoring is used for MAS. "0" means no increase in muscle tone. "5" means affected part(s) rigid in flexion or extension. The validity and reliability of this scoring method in hemiparetic individuals have been shown with different studies.The spasticity values of quadriceps femoris muscle, hip adductor muscles, and gastrocnemius muscles in hemiparetic lower extremities of the participants were recorded. In addition, the total MAS score was determined in the affected lower extremity by summing up all values.
The Single Leg Stance Test | 1 year
  Evaluation of static balance: The Single Leg Stance Test (SLST) from Transitions/Anticipatory Postural Adjustments section, one of the BESTest Balance Evaluation System sub-parameters, was used.While SLST is performed, the patient's stance times on the right and left legs were recorded. During the test, a scoring between 0 and 3 was made according to whether or not the stability of two extremities could be maintained.The highest score a patient could receive was 6. Receiving a high score from four tests indicates that upright position was maintained.
Timed "Get Up & Go" Test | 1 year
  Evaluation of dynamic balance: The Timed "Get Up & Go" Test(TUG) from Stability in Gait section, one of the BESTest Balance Evaluation System sub-parameters, was used.The test started while the patient was sitting on a chair. Three meters from the chair was marked with colored tapes. The person was asked to stand up from chair,walk 3 meters forward,turn 180°,and walk back to the chair and sit on the chair.The completion time of the test was recorded in seconds. A scoring between 0-3 was made according to whether or not the balance is maintained during the test. Getting a high score from the test indicated good balance.
Evaluation of Spatio-Temporal Parameters of Gait | 1 year
  BTS G-Walk Spatio-temporal gait analysis system was used to evaluate gait parameters. Measurements were made in a pre-determined walking area of 10 m.In BTS G-Walk gait analysis system, the results are transferred via Bluetooth to the computer using an analysis port(sensor) connected to L4-L5 or L5-S1 levels of the patient.With the BTS G-Walk system,all important information such as spatio-temporal parameters of gait, general gait kinematics,pelvis, and spine kinematics can be reached.While this system compares the left and right extremities of the person with normal values during gait analysis,it also allows kinematic analysis of the pelvis to be performed in three planes.

SECONDARY OUTCOMES:
Measurement of Joint Range of Motion | 1 year
  Joint Range of Motion (ROM) was measured to determine active and passive joint motion limitation that spasticity can cause in muscle structure and secondarily in joint structure. Active and passive knee flexion-extension and ankle dorsiflexion-plantar flexion ROM were measured using a universal goniometer,whose clinical use is simple and rather practical.

CONTACTS AND LOCATIONS:
Overall Officials: FİLİZ ALTUG, Prof., Study Chair — Pamukkale University; GÜLSÜM TIKAÇ, PT, MSc., Principal Investigator — Pamukkale University; UĞUR CAVLAK, Prof., Study Director — Avrasya University

REFERENCES:
- [Derived] Unal A, Altug F, Tikac G, Cavlak U. Effectiveness of matrix-rhythm therapy on increased muscle tone, balance and gait parameters in stroke survivors: a single-blinded, randomized, controlled clinical trial. Acta Neurol Belg. 2021 Jun;121(3):689-699. doi: 10.1007/s13760-020-01391-6. Epub 2020 Jun 14. PMID 32537732